CLINICAL TRIAL: NCT03539913
Title: Efficacy and Safety of Probiotics in the Treatment of Acute Gastroenteritis in Children
Acronym: SABINA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sb 184
Record Dates: First submitted 2018-05-16; First posted 2018-05-30 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Acute Gastroenteritis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Allocation-blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saccharomyces boulardii (Active Comparator): Floratil, 250 mg sachets, twice daily (1 in the morning and 1 in the evening) during 5 consecutive days.
  Interventions: Biological: Probiotic : Saccharomyces boulardii
- Bacillus clausii (Active Comparator): Enterogermina, 5 ml vials, twice daily (1 in the morning and 1 in the evening) during 5 consecutive days.
  Interventions: Biological: Probiotic : Bacillus clausii

INTERVENTIONS:
Biological: Probiotic : Saccharomyces boulardii — Treatment for 5 days
  Arms: Saccharomyces boulardii
Biological: Probiotic : Bacillus clausii — Treatment for 5 days
  Arms: Bacillus clausii

SUMMARY:
* Primary Objective:

  o To assess the efficacy of the probiotics in reducing the duration of diarrhea in children suffering from acute gastroenteritis.
* Secondary Objectives:

  * To assess the efficacy of the probiotics in improving the frequency and consistency of stools.
  * To assess the efficacy of the probiotics in avoiding recurrence of diarrhea.
  * To assess the efficacy of the probiotics on the disease severity.
  * To assess the safety and tolerability of the studied probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Children of both gender aged between 6 months and 5 years
* Presenting with acute diarrhea (3 or more loose or liquid stools in a 24-hour period) since at least the last 24h but less than 5 days
* Signed informed consent of the legal representatives obtained before any study procedure
* Parents able to fulfill in the stool diary according to the physician's opinion.

Exclusion Criteria:

* Unable to take medication and fluids by mouth
* More than 50% breastfeeding
* Severe malnutrition, defined by a ratio weight/height at/or below -3SD
* Severe dehydration, defined by a need of IV rehydration
* Chronic underlying disease, including but not limited to severe gastrointestinal disorder, immunocompromised condition or systemic infection
* Use of prohibited treatments
* Contra-indications to the studied probiotics

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 317 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-06-09 (Actual)

PRIMARY OUTCOMES:
Time frame in hours up to the time of the last liquid or loose stool as recorded in the stool diary | 5 days
  Time frame in hours up to the time of the last liquid or loose stoll (defined as type 6 or 7 on Bristol Stool Scale) followed by the first 24-hour period with stool consistency improvement (no liquid or loose stool), i.e. cessation of diarrhea as recorded by the parents in the stool diary.

CONTACTS AND LOCATIONS:
Overall Officials: Carine FRANCOIS, Study Director — Biocodex
Locations (8):
- Argentina (8):
  - Instituto Medico, Río Cuarto, Córdoba Province
  - Instituto Medico, San Juan, San Juan Province
  - Instituto Medico, San Miguel de Tucumán, Tucumán Province
  - Consultario Privado 3, CABA
  - Consultorio Privado 1, CABA
  - Consultorio Privado 2, CABA
  - Consultorio Privado 4, CABA
  - Grupo Pediatrico, CABA

REFERENCES:
- [Derived] Altcheh J, Carosella MV, Ceballos A, D'Andrea U, Jofre SM, Marotta C, Mugeri D, Sabbaj L, Soto A, Josse C, Montestruc F, McFarland LV. Randomized, direct comparison study of Saccharomyces boulardii CNCM I-745 versus multi-strained Bacillus clausii probiotics for the treatment of pediatric acute gastroenteritis. Medicine (Baltimore). 2022 Sep 9;101(36):e30500. doi: 10.1097/MD.0000000000030500. PMID 36086703
- [Derived] Collinson S, Deans A, Padua-Zamora A, Gregorio GV, Li C, Dans LF, Allen SJ. Probiotics for treating acute infectious diarrhoea. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD003048. doi: 10.1002/14651858.CD003048.pub4. PMID 33295643